CLINICAL TRIAL: NCT01459198
Title: A Phase I Study of the Safety and Immunogenicity of the Recombinant Live-Attenuated Respiratory Syncytial Virus Vaccine, RSV MEDI ΔM2-2 Lot RSV#002A, Delivered as Nose Drops to Adults 18 to 49 Years of Age, RSV-Seropositive Children 12 to 59 Months of Age, and RSV-Seronegative Infants and Children 6 to 24 Months of Age
Brief Title: Evaluating the Safety and Immune Response to a Respiratory Syncytial Virus (RSV) Vaccine in Adults, RSV-Seropositive Children, and RSV-Seronegative Infants and Children
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CIR 275
Record Dates: First submitted 2011-10-21; First posted 2011-10-25 (Estimated); Last update posted 2015-12-15 (Estimated); Status verified 2015-12

CONDITIONS: Respiratory Syncytial Virus Infections
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Adults: Vaccine (Group 1) (Experimental): Adult participants will receive one dose of the 10^6 RSV MEDI ΔM2-2 vaccine intranasally.
  Interventions: Biological: RSV MEDI ΔM2-2 vaccine
- Seropositive Children: Vaccine (Group 2) (Experimental): Seropositive children will receive one dose of the 10^6 RSV MEDI ΔM2-2 vaccine intranasally.
  Interventions: Biological: RSV MEDI ΔM2-2 vaccine
- Seropositive Children: Placebo Vaccine (Group 2) (Placebo Comparator): Seropositive children will receive one dose of the placebo vaccine intranasally.
  Interventions: Biological: Placebo vaccine
- Seronegative Infants and Children: Vaccine (Group 3) (Experimental): Seronegative infants and children will receive one dose of the 10^5 RSV MEDI ΔM2-2 vaccine intranasally.
  Interventions: Biological: RSV MEDI ΔM2-2 vaccine
- Seronegative Infants and Children: Placebo Vaccine (Group 3) (Placebo Comparator): Seronegative infants and children will receive one dose of the placebo vaccine intranasally.
  Interventions: Biological: Placebo vaccine
- Seronegative Infants and Children: Vaccine (Group 4) (Experimental): Seronegative infants and children will receive one dose of the 10^6 RSV MEDI ΔM2-2 vaccine intranasally.
  Interventions: Biological: RSV MEDI ΔM2-2 vaccine
- Seronegative Infants and Children: Placebo Vaccine (Group 4) (Placebo Comparator): Seronegative infants and children will receive one dose of the placebo vaccine intranasally.
  Interventions: Biological: Placebo vaccine

INTERVENTIONS:
Biological: RSV MEDI ΔM2-2 vaccine — Given intranasally once at a baseline study visit, at a dose of 10^5 or 10^6 plaque-forming units (PFU), depending on study arm.
  Arms: Adults: Vaccine (Group 1); Seronegative Infants and Children: Vaccine (Group 3); Seronegative Infants and Children: Vaccine (Group 4); Seropositive Children: Vaccine (Group 2)
Biological: Placebo vaccine — Given intranasally once at a baseline study visit
  Arms: Seronegative Infants and Children: Placebo Vaccine (Group 3); Seronegative Infants and Children: Placebo Vaccine (Group 4); Seropositive Children: Placebo Vaccine (Group 2)

SUMMARY:
Human respiratory syncytial virus (RSV) is a common cause of upper respiratory tract illnesses as well as more severe lower respiratory illnesses, including bronchiolitis and pneumonia. RSV affects almost all children within the first 2 years of life. This study will evaluate the safety and immune response to the RSV MEDI ΔM2-2 vaccine among adults, RSV-seropositive children, and RSV-seronegative infants and children.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety and immune response of the RSV MEDI ΔM2-2 vaccine in the four groups of participants. The study vaccine will be evaluated in adults, in RSV-seropositive children, and in a dose-ranging study in two groups of RSV-seronegative infants and children.

ELIGIBILITY:
Inclusion Criteria for Adults:

* Adult males and nonpregnant, non-nursing females 18 to 49 years old
* In good health without significant medical illness, physical examination findings, or significant laboratory abnormalities in urinalysis, complete blood count (CBC), alanine aminotransferase (ALT), or creatinine, as determined by a study physician, physician assistant, or nurse practitioner
* Available for the duration of the study
* Willing to participate in the study as evidenced by signing the informed consent document
* Female participants of childbearing potential must have negative urine pregnancy tests and must agree to use effective birth control methods (e.g., birth control pills, diaphragm and foam, condoms with spermicide, Depo-Provera) until 28 days after vaccination

Exclusion Criteria for Adults:

* Pregnant, as determined by a positive urine human chorionic gonadotropin (beta-HCG) test
* Breastfeeding
* Females of childbearing potential who are unwilling to practice effective birth control
* Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, or renal disease by history, physical examination, and/or laboratory studies, including urinalysis
* Behavioral, cognitive, or psychiatric disease that, in the opinion of the investigator, affects the ability of the person to understand and cooperate with the study protocol
* Other condition that, in the opinion of the investigator, would jeopardize the safety or rights of a participant in the study or would render the person unable to comply with the protocol
* Has had medical, occupational, or family problems as a result of alcohol or illicit drug use during the 12 months prior to study entry
* History of a severe allergic reaction or anaphylaxis
* History of splenectomy
* Current diagnosis of asthma within the 2 years prior to study entry
* Positive enzyme-linked immunosorbent assay (ELISA) and confirmatory Western blot tests for HIV-1
* Positive ELISA and confirmatory immunoblot tests for hepatitis C virus (HCV)
* Positive ELISA hepatitis B surface antigen (HBsAg)
* Abnormal urinalysis/urine dip
* Known immunodeficiency syndrome
* Receipt of blood products (including immunoglobulin) within the 3 months prior to study entry
* Current smoker unwilling to stop smoking for the duration of the study
* Previous enrollment in an RSV vaccine study
* Known hypersensitivity to any vaccine component
* Has professional and/or personal responsibilities that involve caring for children younger than 59 months of age or for immunosuppressed individuals
* Systolic blood pressure greater than 140 mm Hg or diastolic blood pressure greater than 90 mm Hg
* Body mass index (BMI) greater than 35

Inclusion Criteria for Seropositive Children:

* Healthy children 12 to 59 months of age, whose parent/guardian understands and signs the study informed consent and agrees to vaccine administration following a detailed explanation of the study
* Seropositive for RSV, defined by serum RSV neutralizing antibody titer greater than 1:40
* Person's history has been reviewed and they have undergone a physical examination indicating that s/he is in good health
* Available for the duration of the study

Exclusion Criteria for Seropositive Children:

* Known or suspected impairment of immunological functions, including maternal history of positive HIV test, receiving immunosuppressive therapy including systemic corticosteroids or bone marrow/solid organ transplant recipients (topical steroids, topical antibiotics, and topical antifungal medications are acceptable)
* Major congenital malformations, including congenital cleft palate, cytogenetic abnormalities, or serious chronic disorders
* Previous immunization with an RSV vaccine
* Previous serious vaccine-associated adverse event (AE) or anaphylactic reaction
* Known hypersensitivity to any vaccine component
* Lung or heart disease, including any wheezing event or reactive airway disease. People with clinically insignificant cardiac abnormalities requiring no treatment may be enrolled. People who had one episode of wheezing or received bronchodilator therapy for a single episode of illness in the first year of life but who have not had any additional wheezing episodes or bronchodilator therapy for at least 12 months may also be enrolled.
* Member of a household that includes an immunocompromised individual or infants younger than 6 months of age, other than a study participant
* Attends day care with infants younger than 6 months of age, and whose parent/guardian is unable or unwilling to suspend daycare for 14 days following immunization. Note: children who attend facilities that separate children by age and minimize opportunities for transmission of virus through direct physical or aerosol contact are acceptable.

Inclusion Criteria for Seronegative Infants and Children:

* Healthy children 6 to 24 months of age whose parents/guardians can understand and sign the informed consent and agree to vaccine administration following detailed explanation of the study
* Seronegative for RSV antibody, defined by serum RSV neutralizing antibody titer less than 1:40 determined within 30 days prior to inoculation
* Person's history has been reviewed and they have undergone a physical examination indicating that s/he is in good health
* Available for the duration of the study

Exclusion Criteria for Seronegative Infants and Children:

* Known or suspected impairment of immunological functions, including maternal history of positive HIV test, receiving immunosuppressive therapy including systemic corticosteroids or bone marrow/solid organ transplant recipients (topical steroids, topical antibiotics, and topical antifungal medications are acceptable)
* Major congenital malformations, including congenital cleft palate, cytogenetic abnormalities, or serious chronic disorders
* Previous immunization with an RSV vaccine
* Previous serious vaccine-associated AE or anaphylactic reaction
* Known hypersensitivity to any vaccine component
* Lung or heart disease, including any wheezing event or reactive airway disease. People with clinically insignificant cardiac abnormalities requiring no treatment may be enrolled. People who had one episode of wheezing or received bronchodilator therapy for a single episode of illness in the first year of life but who have not had any additional wheezing episodes or bronchodilator therapy for at least 12 months may also be enrolled.
* Member of a household that includes an immunocompromised individual or infants younger than 6 months of age, other than a study participant
* Attends day care with infants less than 6 months of age, and whose parent/guardian is unable or unwilling to suspend daycare for 14 days following immunization. Children who attend facilities that separate children by age and minimize opportunities for transmission of virus through direct physical or aerosol contact are acceptable.

Temporary Exclusion Criteria for All Participants:

The following are temporary or self-limiting conditions and, once resolved, the person may be enrolled, if otherwise eligible. If the period of temporary exclusion is more than 56 days for adults or more than 30 days for RSV-seronegative children, the person will need to be rescreened. If the period of temporary exclusion is more than 56 days for RSV-seropositive children, a pre-inoculation serum antibody will need to be collected.

* Fever (adult oral temperature of greater than or equal to 100.4°F [38°C] or pediatric rectal temperature of greater than or equal to 100.4°F [38°C]), or upper respiratory illness (rhinorrhea, cough, or pharyngitis), or nasal congestion significant enough to interfere with successful vaccination, or otitis media
* Has received any killed vaccine or live attenuated rotavirus vaccine within the 2 weeks prior to study entry, any other live vaccine within the 4 weeks prior to study entry, or gamma globulin (or other antibody products) within the 3 months prior to study entry
* Has received another investigational vaccine or investigational drug within 28 days of receiving this investigational RSV vaccine
* Has received antibiotics or systemic or nasal steroid therapy for acute illness within the 3 days prior to vaccination (steroid skin creams or lotions and topical antibiotics or antifungal preparations are permitted)
* Infant or child participant has received salicylate (aspirin) or salicylate-containing products within the 1 month prior to study entry
* Infants born at less than 37 weeks gestation and less than 1 year of age

Ages: 6 Months to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2011-08; Primary Completion 2015-06 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Summarize the frequency of solicited adverse events (AEs) and other AEs | Measured through Day 28 for adults and seropositive children and through Day 56 for seronegative infants and children
List the individual clinical solicited AEs and other AEs, graded by severity. These will be displayed in tabular format and stratified by group. | Measured through Day 28 for adults and seropositive children and through Day 56 for seronegative infants and children
Where appropriate, chi-square or Fisher's exact test will be used to determine significant differences between groups | Measured through Day 28 for adults and seropositive children and through Day 56 for seronegative infants and children

SECONDARY OUTCOMES:
List the peak titer and duration of virus shed by each individual participant. Data will be displayed in tabular format. Mean peak titer and mean duration of shedding will be calculated. | Measured through Day 28 for adults and seropositive children and through Day 56 for seronegative infants and children
List the RSV antibody titer pre- and post-vaccination for each individual participant. Data will be displayed in tabular format. Mean antibody titers will be determined. | Measured through Day 28 for adults and seropositive children and through Day 56 for seronegative infants and children
Determine the infectivity of the vaccine, defined as the proportion of vaccinees who either shed vaccine virus and/or had a fourfold or greater rise in serum antibody titer following vaccination | Measured through Day 28 for adults and seropositive children and through Day 56 for seronegative infants and children
Where appropriate, the Mann-Whitney U test or Tukey-Kramer multiple comparison post-test will be used to determine significant differences between groups | Measured through Day 28 for adults and seropositive children and through Day 56 for seronegative infants and children

CONTACTS AND LOCATIONS:
Overall Officials: Ruth A. Karron, MD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- John Hopkins Center for Immunization Research, Baltimore, Maryland, United States

REFERENCES:
- [Background] Nair H, Nokes DJ, Gessner BD, Dherani M, Madhi SA, Singleton RJ, O'Brien KL, Roca A, Wright PF, Bruce N, Chandran A, Theodoratou E, Sutanto A, Sedyaningsih ER, Ngama M, Munywoki PK, Kartasasmita C, Simoes EA, Rudan I, Weber MW, Campbell H. Global burden of acute lower respiratory infections due to respiratory syncytial virus in young children: a systematic review and meta-analysis. Lancet. 2010 May 1;375(9725):1545-55. doi: 10.1016/S0140-6736(10)60206-1. PMID 20399493
- [Background] Hall CB, Weinberg GA, Iwane MK, Blumkin AK, Edwards KM, Staat MA, Auinger P, Griffin MR, Poehling KA, Erdman D, Grijalva CG, Zhu Y, Szilagyi P. The burden of respiratory syncytial virus infection in young children. N Engl J Med. 2009 Feb 5;360(6):588-98. doi: 10.1056/NEJMoa0804877. PMID 19196675